CLINICAL TRIAL: NCT03154112
Title: Validation of a Novel Oxygen Consumption Measurement Technique in Neonates
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Innovision (Unknown)
Responsible Party: Principal Investigator, John Kheir, Staff Physician, Boston Children's Hospital
Other Study IDs: IRB-P00025365
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Neonatal Respiratory Failure; Congenital Heart Defect
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Measurement of oxygen consumption and caloric expenditure — This study will involve an ~1 hour, single point in time measurement of oxygen consumption, carbon dioxide production, resting energy expenditure, and respiratory quotient using two methods while patients are breathing an FiO2 of 40%. These measurements will be measured using the novel, responsive device and compared with gas collected simultaneously collected from a Douglas bag.

SUMMARY:
The measurement of how much oxygen a baby consumes provides important information about the health of the baby, and of how much energy they are consuming. Currently, there is no device which measures either oxygen consumption, or another variable that depends on oxygen consumption - resting energy expenditure - in neonates or infants. Our group has developed a new device which can attach to any ventilator and measures these two variables with accuracy in the preclinical setting, including in rodents as small as severely preterm infants. The purpose of this study is to compare measurements of oxygen consumption and energy expenditure in neonates using this device and comparing it with a gold standard which is rarely used, a Douglas bag method in which expired gas is collected and later analyzed.

ELIGIBILITY:
Inclusion criteria.

1. Mechanically ventilated neonates and infants (<1 year of age).
2. Inpatients in the cardiac or neonatal intensive care unit at Boston Children's Hospital.
3. Assent of patient's intensive care attending physician, including agreement to place patient on 40% oxygen for up to 60 minutes.
4. Written parental informed consent.

Exclusion criteria.

1. Hemodynamic or respiratory instability.
2. Patients on extracorporeal membrane oxygenation support.
3. Clinically significant tracheo-esophageal fistula
4. Measured endotracheal tube leak >20% (i.e. difference between inspiratory and expiratory tidal volumes)

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients will be selected from inpatients in the neonatal or cardiac intensive care unit who are mechanically ventilated.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Oxygen consumption | 1 hour
Carbon dioxide production | 1 hour
Respiratory quotient | 1 hour
Resting energy expenditure | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nachman E, Clemensen P, Santos K, Cole AR, Polizzotti BD, Hofmann G, Leeman KT, van den Bosch SJ, Kheir JN. A Device for the Quantification of Oxygen Consumption and Caloric Expenditure in the Neonatal Range. Anesth Analg. 2018 Jul;127(1):95-104. doi: 10.1213/ANE.0000000000003308. PMID 29505450

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT03154112/Prot_SAP_000.pdf